CLINICAL TRIAL: NCT01200550
Title: An Epidemiological, Observational Study to Describe Symptom Control and Impact on Daily Life in Patients With Gastroesophageal Reflux Disease (GERD)
Brief Title: The Study to Describe Symptom Control and Impact on Daily Life in Gastroesophageal Reflux Disease (GERD) Patients
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-GBA-DUM-2010/1
Record Dates: First submitted 2010-09-07; First posted 2010-09-13 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gastroesophageal reflux disease; GERD Impact Scale
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
The purpose of this study is to evaluate symptoms control and impact on daily life from patients perspective using specific GERD Impact Scale(GIS) questionnaire. The another objective is to obtain local epidemiological data for Bosnia and Herzegovina regarding GERD treatment in primary care.

ELIGIBILITY:
Inclusion Criteria:

* Patients previously diagnosed with GERD (disease duration =3 years) or newly diagnosed patients that are currently not treated with proton pump inhibitor, for whom specialist or General Practionaire (GP) have previously decided to initiate or change treatment for GERD; Patients should be treated for GERD according to current practice

Exclusion Criteria:

* Females of childbearing potential should not be pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients previously diagnosed with GERD (disease duration =3 years) or newly diagnosed patients that are currently not treted with proton pump inhibitors, for whom GP or specialist (in primary care unit) have previosly decided to initiate or change treatment for GERD.
Sampling Method: Probability Sample
Enrollment: 1233 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Epidemiological data: To assess frequency and severity of typical GERD symptoms in newly diagnosed GERD patients and GERD patients with disease duration =3 years | Maximum of 14 weeks, with 3 visits in total
Epidemiological data: To assess frequency and severity of typical GERD symptoms in newly diagnosed GERD patients and GERD patients with disease duration =3 years | Visit 1 (enrolment)
Epidemiological data: To assess frequency and severity of typical GERD symptoms in newly diagnosed GERD patients and GERD patients with disease duration =3 years | Visit 2 (4-6 weeks after Visit 1)
Epidemiological data: To assess frequency and severity of typical GERD symptoms in newly diagnosed GERD patients and GERD patients with disease duration =3 years | Visit 3 (8-14 weeks after Visit 1).

SECONDARY OUTCOMES:
The evaluation of GERD Impact Scale (GIS questionnaire) as a useful tool for initial and long term management of GERD patients | Maximum of 14 weeks, with 3 visits in total: Visit 1 (enrolment), Visit 2 (4-6 weeks after Visit 1) and Visit 3 (8-14 weeks after Visit 1).

CONTACTS AND LOCATIONS:
Overall Officials: Srdjan Gornjakovic, MD, PhD, Principal Investigator — Clinical Center University of Sarajevo; Department of Gastrenterology and HepatologySarajevo
Locations (23):
- Bosnia and Herzegovina (23):
  - Research Site, Banja Luka
  - Research Site, Bijeljina
  - Research Site, Derventa
  - Research Site, Doboj
  - Research Site, Gračanica
  - Research Site, Gradačac
  - Research Site, Gradiška
  - Research Site, Hadžići
  - Research Site, Jelah
  - Research Site, Laktaši
  - Research Site, Lukavac
  - Research Site, Lukavica
  - Research Site, Matuzići
  - Research Site, Mostar
  - Research Site, Pale
  - Research Site, Prijedor
  - Research Site, Sarajevo
  - Research Site, Trn
  - Research Site, Tuzla
  - Research Site, Visoko
  - Research Site, Vogošća
  - Research Site, Zalužani
  - Research Site, Živinice